CLINICAL TRIAL: NCT03167294
Title: PROCEPT AQUABEAM Study for the Treatment of Benign Prostatic Hyperplasia (ABS)
Brief Title: AQUABEAM India Study for the Treatment of Benign Prostatic Hyperplasia
Acronym: ABS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PROCEPT BioRobotics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TP0032
Record Dates: First submitted 2014-12-11; First posted 2017-05-25 (Actual); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Benign Prostatic Hyperplasia
Keywords: Aquablation; AQUABEAM; BPH; LUTS
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm (Other): AquaBeam System for resection and removal of prostatic tissue in males suffering from BPH
  Interventions: Device: AquaBeam System

INTERVENTIONS:
Device: AquaBeam System — Aquablation

SUMMARY:
Single-arm prospective, interventional clinical trial. Results will be compared to a historical control in the treatment of benign prostatic hyperplasia

ELIGIBILITY:
Inclusion Criteria:

* Male
* 50 - 80 years
* Moderate to severe BPH
* Subjects who have failed standard medical therapy

Exclusion Criteria:

* Size and width of prostate
* Medical condition or co-morbidities where BPH intervention would be contraindicated

Ages: 50 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2014-12-14 (Actual); Primary Completion 2016-06-30 (Actual); Study Completion 2017-04-27 (Actual)

PRIMARY OUTCOMES:
Primary Device Performance Endpoint | 6 months
  The primary device performance endpoint is completion of the intended surgical procedure.
Primary Safety Endpoint of the study is the perioperative complication rate. | 6 months
  The primary safety endpoint of the study is the perioperative complication rate

CONTACTS AND LOCATIONS:
Overall Officials: Ravindra Sabnis, Principal Investigator — Chairman, department of Urology Muljibhai Patel Urological Hospital
Locations (1):
- Muljibhai Patel Urological Hospital, Nadiād, Gujarat, India